CLINICAL TRIAL: NCT06078020
Title: PLatform Study for INTracerebral Haemorrhage (PLINTH): Community-based Feasibility Study
Acronym: PLINTH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of the West of Scotland (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: AC23101; HIPS/22/36 (Other Grant/Funding Number: Chief Scientist Office of the Scottish Government); 325272 (Other: Integrated Research Application System)
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Hemorrhage
Keywords: Platform study; Randomised controlled trial; Feasibility study
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Semi-structured interview to assess understanding and acceptability at 3+/-2 and 14+/-7 days after consent

SUMMARY:
The goal of this observational study is to answer three uncertainties about the design of a platform study for adults with stroke due to intracerebral haemorrhage.

The main things the investigators aim to find out are:

* The acceptability of a platform trial and its comparisons to brain haemorrhage survivors or their carers, and their clinicians.
* Estimates of eligibility, willingness to participate, diversity, representativeness, adherence, retention, data completion, and event rates of intermediate and clinical outcomes over time for each comparison.
* The most efficient platform trial design considering the findings of this feasibility study.

Participants, or their welfare guardian, welfare attorney, or nearest relative will:

* Watch a video informing them about the study
* Read written information about the study
* Provide informed consent
* Permit collection of demographic and clinical details
* Provide information in interviews at ~3 and ~14 days after the onset of the stroke

DETAILED DESCRIPTION:
Background: Clinical trials have not found a treatment that works specifically for stroke caused by bleeding in the brain, known as intracerebral haemorrhage (ICH for short). Most clinical trials have studied one treatment at a time and included only 1 in 10 people with ICH. That's why each clinical trial recruited only 77 participants on average. A PLatform trial for INTracerebral Haemorrhage (PLINTH) will change this by investigating several treatments and giving everyone with ICH an opportunity to take part.

Aim: The investigators intend PLINTH to be large, inclusive, efficient and assess several treatments for ICH. First, a feasibility study is needed to work out whether PLINTH can succeed.

Methods: The investigators will find people recently diagnosed with ICH in Lothian and Lanarkshire and invite them to take part in a feasibility study. The investigators will provide them with personalised information using Tailored Talks. The investigators will find out if PLINTH is acceptable to people with ICH, carers, and doctors. The investigators will use data that are collected routinely to follow participants' progress. Characteristics and outcomes of participants will help design PLINTH.

Patient & public involvement: The investigators asked ICH survivors about PLINTH: 92% strongly agreed that working out how to do a platform study to find treatments for ICH is a priority. An ICH survivor is in the study team.

Dissemination: The investigators will produce easy access reports and share them with people with ICH, carers, healthcare professionals, and the public in their preferred format (printed, email, social media, and on the Research to Understand Stroke due to Haemorrhage website [http://www.RUSH.ed.ac.uk]).

ELIGIBILITY:
Inclusion Criteria:

* People aged ≥18 years at the time of diagnosis with symptomatic stroke due to first-ever or recurrent spontaneous (non-traumatic) ICH, most likely to be due to cerebral small vessel disease, confirmed by brain imaging between 1 October 2023 and 30 June 2025 inclusive
* One or more management uncertainties exist about the patient's management according to the patient/nearest relative and their responsible clinician
* Patient or their nearest relative can be approached for consent to participation in this feasibility study with the aid of simple information delivered by Tailored Talks
* Residential postcode in the National Health Service (NHS) Lothian or NHS Lanarkshire regions of Scotland

Exclusion Criteria:

* People aged <18 years at the time of ICH diagnosis
* Exclusively extra-axial intracranial haemorrhage or ICH definitely attributable to a macrovascular cause (e.g. aneurysm, arteriovenous malformation, cavernoma, cerebral venous sinus thrombosis), tumour, trauma or haemorrhagic transformation of an ischaemic stroke
* Responsible clinician deems it inappropriate to approach the patient or their nearest relative (e.g. death appears imminent)
* Mental incapacity and no nearest relative, welfare attorney or welfare guardian available at the time of approach
* Patient died before approached for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with stroke due to intracerebral haemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 21 months
  The frequency of people with incident ICH for whom there is at least one management uncertainty about ICH, with consent to participate in this feasibility study, and willingness to consider participating in a future PLINTH

SECONDARY OUTCOMES:
Estimates required for the design of an inclusive and representative future PLINTH | 21 months
  Demographic and clinical characteristics of people incident with ICH who would participate in a future PLINTH
Feasibility of the consent process | 21 months
  Acceptability to participants of an electronic approach to providing personalised information about their care and shared decision making about potential eligibility for recruitment to a future PLINTH (video abstract and Tailored Talks)

CONTACTS AND LOCATIONS:
Overall Officials: Rustam AS Salman, MA PhD FRCPE, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - The Royal Infirmary of Edinburgh, Edinburgh, City Of Edinburgh
  - University Hospital Monklands, Airdrie, Lanarkshire

IPD SHARING:
Plan to Share IPD: Yes
Once the data retention period is over, study data will be de-identified and archived in the University of Edinburgh's secure DataShare (https://datashare.ed.ac.uk/), an open access repository.
Supporting Information: Study Protocol, ICF
Time Frame: One year after completion of the study
Access Criteria: Data collected or generated by the study may be transferred to any external individuals or organisations outside of the Sponsoring organisation(s) under a defined data sharing agreement.
URL: https://www.ed.ac.uk/plinth

REFERENCES:
- See also: Study website — https://www.ed.ac.uk/plinth